CLINICAL TRIAL: NCT01407289
Title: An Open, Single-centre, Controlled Trial to Investigate the Efficacy and Usability of Published Best Practice to Control Glycaemia in Hospitalised Patients With Type 2 Diabetes
Brief Title: A Trial to Investigate Efficacy and Usability of Published Best Practice to Control Glycaemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Pieber Thomas, MD, MD, Prof. of Medicine, Medical University of Graz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ClinDiab-02
Record Dates: First submitted 2011-07-19; First posted 2011-08-02 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; Insulin Glargine

ARMS (2):
- Insulin titration protocol (Experimental): Patients in care at the Division of Endocrinology will be treated by enhanced version of published best paper based practice insulin titration protocol to control glycaemia in hospitalised patients with type 2 diabetes.
  Interventions: Drug: Insulin Aspart, Insulin Glargine
- Standard care (No Intervention): Patients in care of the Division of Cardiology will be treated using antihyperglycaemic therapy according to standard care.

INTERVENTIONS:
Drug: Insulin Aspart, Insulin Glargine — The Intervention is a paper based protocol, which provides suggestions for new insulin doses (basal-bolus regime).
  Arms: Insulin titration protocol

SUMMARY:
The purpose of the study is to compare the efficacy of enhanced published best practice paper-based insulin titration protocol for glycaemic control in hospitalised patients with type 2 diabetes for the length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Blood glucose in the range between 140 - 400 mg/dl
* Expected stay ≥ 48 hours

Exclusion Criteria:

* Hyperglycemia without known history of type 2 diabetes mellitus
* Impaired renal function (serum creatinine ≥3.0mg/dL)
* Clinically relevant hepatic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Mean blood glucose | duration of hospital stay (48 hours - maximum three weeks)
  Mean blood glucose over 24 hours

SECONDARY OUTCOMES:
Number of glucose measurements in hyperglycaemic ranges | duration of hospital stay (48 hours - maximum three weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pieber, MD, Principal Investigator — Division of Endocrinology and Metabolism, Department of Internal Medicine Medical University of Graz
Locations (1):
- Medical University of Graz, Division of Internal Medicine, Department of Endocrinology and Metabolism/ Cardiology, Graz, Austria

REFERENCES:
- [Derived] Donsa K, Beck P, Holl B, Mader JK, Schaupp L, Plank J, Neubauer KM, Baumgartner C, Pieber TR. Impact of errors in paper-based and computerized diabetes management with decision support for hospitalized patients with type 2 diabetes. A post-hoc analysis of a before and after study. Int J Med Inform. 2016 Jun;90:58-67. doi: 10.1016/j.ijmedinf.2016.03.007. Epub 2016 Mar 23. PMID 27103198
- [Derived] Schaupp L, Donsa K, Neubauer KM, Mader JK, Aberer F, Holl B, Spat S, Augustin T, Beck P, Pieber TR, Plank J. Taking a Closer Look--Continuous Glucose Monitoring in Non-Critically Ill Hospitalized Patients with Type 2 Diabetes Mellitus Under Basal-Bolus Insulin Therapy. Diabetes Technol Ther. 2015 Sep;17(9):611-8. doi: 10.1089/dia.2014.0343. Epub 2015 Apr 30. PMID 25927357